CLINICAL TRIAL: NCT02808364
Title: Personalized Cellular Vaccine Therapy in Treating Patients With Recurrent Glioblastoma (PerCellVac2)
Brief Title: Personalized Cellular Vaccine for Recurrent Glioblastoma (PERCELLVAC2)
Acronym: PerCellVac2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong 999 Brain Hospital (Other)
Collaborators: Beijing Tricision Biotherapeutics Inc (Industry); Zhuhai Trinomab Pharmaceutical Co., Ltd. (Industry); Jinan University Guangzhou (Other)
Responsible Party: Principal Investigator, Jian Zhang, Vice President of the hospital and Chief Physician, Guangdong 999 Brain Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ag-mRNA-Cell-999brain
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Glioblastoma
Keywords: Recurrent glioblastoma; DC vaccine; tumor antigen; personalized vaccine
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Personalized cellular vaccine (Experimental): Subjects will undergo tumor resection. They will receive biweekly cellular vaccines consisting of mRNA tumor antigen pulsed autologous DCs.
  Interventions: Biological: Personalized cellular vaccine

INTERVENTIONS:
Biological: Personalized cellular vaccine — Patients with recurrent glioblastoma will undergo tumor resection and receive tumor antigen pulsed cellular vaccines.
  Other Names: Tumor antigen pulsed DC autologous cellular vaccine

SUMMARY:
The treatment option for recurrent glioblastoma is limited. Immune cell based therapy for glioblastoma has shown some efficacy. This study is designed to perform a personalized clinical trial by first analyzing the expression of tumor associated antigens in patients with recurrent glioblastoma and then immunizing the patients with personalized antigen pulsed DCs. Immune responses to the immunized antigens will be monitored. Safety and efficacy will be observed in this study.

DETAILED DESCRIPTION:
This is an open label, single-arm, single-institution, Phase I study designed to investigate the safety and efficacy of personalized cellular vaccines for patients with recurrent glioblastoma (GBM). Recurrent GBM patients will undergo tumor resection. The tumors will be analyzed for the expression of a panel of glioma-associated antigens and immune-related genes. Patients will undergo leukapheresis to collect mononuclear cells for DC generation. Based on the expression profiles of tumor-associated antigens, in vitro transcribed mRNA will be generated to pulse autologous DCs. Patients will be conditioned with immune adjuvants before and during immunization. Patients will receive biweekly vaccines. The antitumor specific T cell responses will be measured. Safety and efficacy will be monitored. The objective is to assess the safety of the personalized cellular vaccines and T cell responses. The efficacy of the vaccines will be evaluated using iRANO criteria, progression-free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent glioblastoma grade IV
* Patients at the age of 18-65.
* Patients undergo tumor resection.
* Patients with Karnofsky scores > or =70
* Patients with normal range of hematologic and metabolic test results.
* Patients must have no corticosteroids treatment at least one week before vaccination.
* Patients capable of understanding the study and signed informed consent.

Exclusion Criteria:

* Breast feeding females.
* Pregnant women.
* Infectious diseases HIV, HBV, HCV
* Documented immunodeficiency
* Documented autoimmune disease
* Any serious or uncontrolled medical or psychiatric conditions, for example, severe pulmonary, cardiac or other systemic disease.
* Patient inability to participate as determined by PI discretion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events and severe adverse events (safety and tolerability) | 3 years since the beginning of the first vaccine
  Incidence of adverse events and severe adverse events to measure safety and tolerability of mRNA-TAA pulsed autologous DC, allogeneic PBMCs and autologous tumor cellular vaccines.

SECONDARY OUTCOMES:
Antitumor antigen specific T cell response | 4 weeks after the last vaccine
  The frequency of the peripheral CD8+ and CD4+ T cell response to the vaccine will be measured.
Progression-free survival | 12 months since the beginning of the first vaccine
  Progression-free survival will be monitored for 1 year.
Overall survival | 3 years since the beginning of the first vaccine
  Overall survival will be monitored for 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, M.D., Principal Investigator — Guangdong 999 Brain Hospital
Locations (1):
- Guangdong 999 Brain Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wang QT, Nie Y, Sun SN, Lin T, Han RJ, Jiang J, Li Z, Li JQ, Xiao YP, Fan YY, Yuan XH, Zhang H, Zhao BB, Zeng M, Li SY, Liao HX, Zhang J, He YW. Tumor-associated antigen-based personalized dendritic cell vaccine in solid tumor patients. Cancer Immunol Immunother. 2020 Jul;69(7):1375-1387. doi: 10.1007/s00262-020-02496-w. Epub 2020 Feb 20. PMID 32078016
- See also: Clinical trial results — https://pubmed.ncbi.nlm.nih.gov/32078016/